CLINICAL TRIAL: NCT07398716
Title: Intraoperative Assessment of Distal Resection Margins Using Frozen Section in Mid and Low Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Nurettin Şahin, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOFS-DM
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer
Keywords: frozen section; Distal resection margin; Low rectal cancer; Mid rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Frozen Sections

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, two-arm, parallel-group interventional study comparing intraoperative frozen section assessment of distal resection margins versus standard surgery in mid and low rectal cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Frozen Section Group (Experimental): Patients undergo total mesorectal excision followed by intraoperative colonoscopy.
  After specimen removal, distal resection margins are assessed using intraoperative frozen section by an expert pathologist.
  Additional resection is performed if margins are positive or less than 1 cm. Abdominoperineal resection is performed if a safe margin cannot be achieved.
  Interventions: Procedure: Intraoperative Frozen Section Assessment
- Control Group (Active Comparator): Patients undergo total mesorectal excision followed by intraoperative colonoscopy.
  Resection is performed 2 cm distal to the tumor using a stapler, and anastomosis is completed without intraoperative frozen section assessment.
  Interventions: Procedure: Standard Surgery Without Frozen Section

INTERVENTIONS:
Procedure: Intraoperative Frozen Section Assessment — Intraoperative pathological evaluation of distal resection margins using frozen section to guide surgical decision-making.
  Arms: Intraoperative Frozen Section Group
Procedure: Standard Surgery Without Frozen Section — Standard surgical resection without intraoperative frozen section assessment of distal margins.
  Arms: Control Group

SUMMARY:
This study aims to improve the safety of distal surgical margins in patients with middle and low rectal cancer who receive neoadjuvant radiotherapy. Although magnetic resonance imaging and colonoscopic evaluation after neoadjuvant radiotherapy may suggest complete or near-complete tumor regression, residual tumor cells can still be present in the submucosal and muscular layers of the rectal wall. This may increase the risk of inadequate surgical margins and local recurrence.

In this study, patients with middle and low rectal cancer who are scheduled for surgery after neoadjuvant radiotherapy will be randomized into two groups. In the frozen section group, intraoperative frozen section analysis of the resection specimen will be performed immediately after specimen removal to assess the distal resection margin, and the surgical procedure will be guided according to the frozen section results. In the control group, standard surgical resection will be performed without intraoperative frozen section evaluation.

Pathological findings, distal margin status, operative time, tumor stage, and recurrence during follow-up will be compared between the two groups to evaluate the impact of intraoperative frozen section analysis on surgical margin safety and oncological outcomes.

DETAILED DESCRIPTION:
Middle and low rectal cancers often show a good response to neoadjuvant radiotherapy or chemoradiotherapy. However, despite apparent tumor regression or disappearance on preoperative magnetic resonance imaging and intraoperative colonoscopic evaluation, residual tumor cells may persist within the submucosal or muscular layers of the rectal wall. This residual disease may not be detected by mucosal inspection alone and may lead to inadequate distal resection margins, increasing the risk of local recurrence or the need for more radical surgery.

The primary aim of this study is to evaluate whether intraoperative frozen section analysis of the distal resection margin improves surgical margin safety in patients with middle and low rectal cancer undergoing surgery after neoadjuvant radiotherapy.

This is a prospective, randomized clinical study conducted at Bakırköy Dr. Sadi Konuk Training and Research Hospital. Patients diagnosed with middle or low rectal adenocarcinoma (stage I-III) who have undergone short-course or long-course neoadjuvant radiotherapy and have been discussed in a multidisciplinary oncology council will be included. Following restaging with pelvic magnetic resonance imaging, patients deemed suitable for surgical treatment will be enrolled.

Eligible patients will be randomized into two groups using a sealed-envelope method. All patients will undergo total mesorectal excision according to standard oncologic principles. Immediately before rectal transection, intraoperative colonoscopy will be performed in all patients, and rectal transection will be planned at 2 cm distal to the tumor site identified during colonoscopy using an endoscopic linear stapler.

In the frozen section group, after specimen removal, the resection specimen will be immediately evaluated by an experienced gastrointestinal pathologist using intraoperative frozen section analysis. A distal margin of at least 1 cm will be considered oncologically safe. If the distal margin is found to be positive or closer than 1 cm, further rectal resection will be performed until a safe margin is achieved. If a safe distal margin cannot be obtained despite additional resection, abdominoperineal resection will be performed.

In the control group, after specimen removal, anastomosis will be performed without intraoperative frozen section analysis, and the operation will be completed according to standard surgical practice.

At the end of surgery, all specimens from both groups will undergo routine formalin-fixed pathological examination, including tumor staging and assessment of distal and circumferential resection margins.

Patient demographics, operative time, pathological tumor stage, distal margin status, need for additional resection or abdominoperineal resection, and recurrence during follow-up will be recorded and compared between the two groups.

The results of this study aim to determine whether intraoperative frozen section analysis contributes to safer distal surgical margins and improved oncological decision-making in the surgical treatment of middle and low rectal cancer following neoadjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mid or low rectal cancer (Stage I-III)
* Patients who have received short-course or long-course neoadjuvant radiotherapy
* Patients evaluated and approved for surgery by a multidisciplinary oncology board
* Patients scheduled for total mesorectal excision (TME)
* Age ≥ 18 years
* Patients who provide written informed consent

Exclusion Criteria:

* Stage IV rectal cancer
* Upper rectal tumors
* Patients undergoing emergency surgery
* Patients planned for local excision or palliative surgery
* Patients with distant metastasis
* Patients with a history of previous rectal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of Negative Distal Resection Margin (R0) | During surgery
  Patients who obtained a negative result at the distal resection margin (defined as a tumor-free margin of at least 1 cm) according to intraoperative frozen section examination.

SECONDARY OUTCOMES:
Need for Additional Resection or Conversion to Abdominoperineal Resection (APR) | During surgery
  The proportion of patients requiring additional distal rectal resection or conversion to abdominoperineal resection due to positive or insufficient distal resection margins.
Local Recurrence Rate | During postoperative follow-up (12- 24 months)
  The incidence of local tumor recurrence during postoperative follow-up, confirmed by imaging, endoscopy, or pathological evaluation.
Operative Time | During surgery
  Total duration of the surgical procedure measured from skin incision to completion of wound closure.

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin Sahin, MD, Principal Investigator — Bakırköy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Bakırköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the study is a single-center trial and data sharing was not included in the original ethics committee approval. De-identified aggregate data may be available upon reasonable request to the corresponding investigator

REFERENCES:
- [Result] Gomes RM, Bhandare M, Desouza A, Bal M, Saklani AP. Role of intraoperative frozen section for assessing distal resection margin after anterior resection. Int J Colorectal Dis. 2015 Aug;30(8):1081-9. doi: 10.1007/s00384-015-2244-4. Epub 2015 May 16. PMID 25982468
- [Result] Khoury W, Abboud W, Hershkovitz D, Duek SD. Frozen section examination may facilitate reconstructive surgery for mid and low rectal cancer. J Surg Oncol. 2014 Dec;110(8):997-1001. doi: 10.1002/jso.23758. Epub 2014 Sep 2. PMID 25183166